CLINICAL TRIAL: NCT00680212
Title: Phase 2 Study of VITAMIN A EQUIVALENCE OF PLANT CAROTENOIDS IN CHILDREN
Brief Title: Vitamin A Equivalence of Plant Carotenoids in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Guangwen Tang, Tufts University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 8458; R01DK060021 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Vitamin A Deficiency
Keywords: dietary beta-carotene; vitamin A status; intrinsically labeled plant foods
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): dietary carotenoids
  Interventions: Dietary Supplement: dietary carotenoids; Dietary Supplement: spinach, rice, and synthetic beta-carotene

INTERVENTIONS:
Dietary Supplement: dietary carotenoids — spinach containing 1 - 2 mg beta-carotene rice containing 0.5 mg beta-carotene synthetic beta-carotene 0.5 mg oil capsule
Dietary Supplement: spinach, rice, and synthetic beta-carotene — spinach containing 1 - 2 mg beta-carotene rice containing 0.5 mg beta-carotene synthetic beta-carotene, 0.5 mg oil dose
  Other Names: dietary carotenoids

SUMMARY:
Our objectives will be to test the following hypotheses and to make the following determinations: (1) The absorption and bio-conversion of provitamin A carotenes taken by children are different between spinach, Golden Rice, and ß-C in oil capsules. (2) The absorption of provitamin A carotenes and their bioconversion to vitamin A are different in children with or without adequate vitamin A nutrition. (3) To define the vitamin A equivalence(s) of dietary spinach, Golden Rice, and a ß-C in oil dose by using an isotope reference method in children with or without adequate vitamin A nutrition and to compare those values with values derived from model based compartmental analysis. (4) To determine the number and time of blood samples needed for future studies in various field settings on the retinol equivalence of a large number of plant sources.

DETAILED DESCRIPTION:
This project is to determine the vitamin A value (equivalence) of dietary provitamin A carotenes from spinach, Golden Rice, and pure ß-carotene (ß-C) in oil. These experiments will be conducted in children (ages 6-8) with/without adequate (marginal deficiency) vitamin A nutrition. As plant provitamin A carotenoids are a major and safe vitamin A source for a vast population in the world, it is essential to determine the efficiency of provitamin A carotenoid (mainly ß-C) conversion to vitamin A. By introducing ß-C into rice endosperm, Golden Rice may directly benefit consumers by providing vitamin A nutrition. Our investigation uses hydroponically grown, deca-deuterium labeled spinach and Golden Rice, synthetic ß-C-d10 and a vitamin A isotope reference, C13 labeled retinyl acetate (13C10-RAc), to evaluate the bioavailability and the bioconversion of plant provitamin A carotenes to retinol as compared with ß-C in oil capsules in vivo.

Seventy-two children each will take two meals, breakfast containing 13C10-RAc dose (0.5mg in 0.2g oil capsule) and lunch containing spinach containing 1 mg ß-C (along with white rice), or Golden Rice containing 0.5mg ß-C (along with light colored vegetables), or ß-C oil capsules containing 0.5 mg ß-C in 0.2g oil (along with white rice and light colored vegetables) on the first day of the study. Blood samples will be collected at 1 3, 7, 14, and 21 days after the study doses.

The enrichment of labeled ß-C and labeled retinol in human circulation will be determined using advanced liquid chromatography / mass spectrometry and gas chromatography / mass spectrometry. Through the applications of these novel technologies, we will be able to determine the relative biological activities of endogenous carotenoids; that is, the vitamin A value of spinach, Golden Rice, and ß-C in oil capsules for children with/without vitamin A malnutrition.

This study will be of importance in planning vitamin A deficiency prevention strategies and also will provide useful information regarding the potential efficacy of a bioengineered crop to provide vitamin A nutrition.

ELIGIBILITY:
Inclusion Criteria:

* healthy children

Exclusion Criteria:

* food allergy
* parasitic infection

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
conversion efficiency of b-C to retinol | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Guangwen Tang, Ph. D, Principal Investigator — Tufts University
Locations (1):
- USDA Human Nutrition Research Center on Aging, Tufts Uni., Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tang G, Hu Y, Yin SA, Wang Y, Dallal GE, Grusak MA, Russell RM. beta-Carotene in Golden Rice is as good as beta-carotene in oil at providing vitamin A to children. Am J Clin Nutr. 2012 Sep;96(3):658-64. doi: 10.3945/ajcn.111.030775. Epub 2012 Aug 1. PMID 22854406 (Retraction: PMID 26224301 Am J Clin Nutr. 2015 Sep;102(3):715)